CLINICAL TRIAL: NCT00362063
Title: Effects of Growth Hormone on Glucose and Protein Metabolism in Children With Growth Hormone Deficiency
Brief Title: 304-C03/L3301n: Effects of Growth Hormone on Glucose and Protein Metabolism in Children With Growth Hormone Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Luisa M. Rodriguez, Principal Investigator, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-14859
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Growth Hormone Deficiency
Keywords: growth hormone
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone; Human Growth Hormone

ARMS (2):
- growth hormone (Experimental): children with proven growth hormone deficiency
  Interventions: Drug: growth hormone (Nutropin)
- healthy controls (No Intervention): No growth hormone is given

INTERVENTIONS:
Drug: growth hormone (Nutropin) — growth hormone (Nutropin), 0.3mg/kg/week administered subcutaneously daily.
  Arms: growth hormone

SUMMARY:
The purpose of the proposed study is to investigate the effects of rhGH treatment on glucose, protein and fat metabolism in GHD children. Specifically, the investigators will measure the rates of glucose production, gluconeogenesis, glycogenolysis, insulin sensitivity and glucagon response before and after treatment with rhGH. In addition, the investigators will study changes in protein and fat metabolism pre and post rhGH therapy in children with GHD. The findings in the GHD children will be compared to those of a control group of age and sex matched healthy children.

Hypotheses: H1- The fraction of glucose derived from gluconeogenesis is decreased and that from glycogenolysis is increased in the post-absorptive state in untreated GHD children when compared to healthy children. H2- Treatment with rhGH will not change the overall glucose turnover but will normalize the abnormal partitioning of gluconeogenesis and glycogenolysis in GHD children. H3- GH replacement will reduce urea production and increase estimates of protein synthesis, thus optimizing the availability of amino acids for growth. H4- Untreated children with GHD after an overnight fast will have an increased glucagon challenge response that will decrease after 8 weeks of treatment with rhGH.

Specific Aims: In healthy and newly diagnosed GHD children the investigators will: 1. Measure the Glucose Production Rate (GPR) 2. Determine the fraction of glucose derived from gluconeogenesis and glycogenolysis 3. Estimate insulin sensitivity 4. Measure proteolysis and protein oxidation 5. Determine glucagon challenge response after an overnight fast. The above-mentioned parameters will be re-evaluated in the children with GHD after 8 weeks of rhGH therapy.

DETAILED DESCRIPTION:
Children with growth hormone deficiency (GHD) have increased insulin sensitivity and may present with hypoglycemia during infancy. Treatment with recombinant human growth hormone (rhGH) reduces the risk for hypoglycemia and decreases insulin sensitivity. The investigators hypothesize, that GHD causes a decrease in the fraction of glucose derived form gluconeogenesis and conversely glycogenolysis and insulin sensitivity will be increased, when GHD children are compared to healthy controls. The investigators anticipate that total glucose production will be unaffected by rhGH therapy. Therefore, the GDH subjects treated with rhGH for 8 weeks will have an increase in the fraction of glucose derived form gluconeogenesis and a decrease in that form glycogenolysis and decreased insulin sensitivity. To test this hypothesis, 10 healthy and 10 GHD children will be studied using the stable isotope [U-13C] glucose and Mass Isotopes Distribution Analysis (MIDA). The investigators will be specifically measuring the rate of glucose production, gluconeogenesis, glycogenolysis, insulin sensitivity and glucagon response after an overnight fast. In addition, the investigators will measure changes in protein oxidation, proteolysis and fat metabolism using the stable isotopes [15N2] urea, [1-13C] leucine and concentrations of free fatty acids and b-hydroxybutyrate. The GHD group will be studied at the time of diagnosis and after 8 weeks of rhGH.

ELIGIBILITY:
Inclusion Criteria:

The study population will consist of children with newly diagnosed growth hormone deficiency (GHD), between the ages of 1-17 years. The clinical evidence will be provided by one or more of the following criteria: delayed bone age, growth deceleration, short stature (more than 2 SD bellow the mean for the subject's age) and/ or height more than1.5 SD below the predicted mid-parental height. The biochemical diagnosis of GHD will be established by an abnormal growth hormone stimulation test and low IGF-1 and IGFBP-3 (growth factors). The growth hormone stimulation test will be performed following the standard Endocrinology Clinic protocol. The growth hormone stimulation test is considered the "gold standard" to diagnose Growth Hormone Deficiency. This test is part of the standard clinical practice to diagnosed GHD. An abnormal test is defined as a post stimulation Growth Hormone level less than10 ng/mL.

The control group will include healthy children between the ages of 1-17 years, not taking any medication with a normal weight for height and growth factors (IGF-1 and IGFBP-3)."

Exclusion Criteria:

The exclusion criteria will include for both groups age less than 1 or more than 17 y/o, evidence of anemia (hemoglobin less tan 12 mg/dl), the use of medications that can directly impact blood sugar (steroids, oral contraceptives etc), history or proof of chemical abuse, lack of supportive family environment, allergies to local anesthetics and elevated liver enzymes. The GHD children will have a head MRI, and children with evidence of tumors or space occupying lesions will be excluded. GHD subjects with adrenal insufficiency and or hypothyroidism. will not be considered for the study.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Glucose Production rate,Gluconeogenesis, glycogenolysis. | 13 hours fasting

SECONDARY OUTCOMES:
Insulin resistance | 13 hours fasting
Proteolysis | 13 hours fasting
Glucagon response | for 2hrs after glucagon administration

CONTACTS AND LOCATIONS:
Overall Officials: Luisa M Rodriguez, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States